CLINICAL TRIAL: NCT06543056
Title: An Open-label, Single-arm Phase 2 Study of ES014 in Subjects With Advanced Solid Tumors
Brief Title: A Study of ES014 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Elpiscience (Suzhou) Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES014-IIT-01
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
Keywords: ES014; CD39/TGF-β; Advanced Solid Tumor; Phase II
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ES014 (Experimental): ES014 will be administered in patients with advanced solid tumors.
  Interventions: Drug: ES014

INTERVENTIONS:
Drug: ES014 — ES014 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 24 months.
  Other Names: ES014 for Injection

SUMMARY:
OVERALL DESIGN: This study is an open-label, single-center, single-arm phase 2 clinical study designed to evaluate the efficacy, safety, and tolerability of ES014 in adults with advanced solid tumors. Adult patients with unresectable locally advanced or metastatic solid tumors will be enrolled in this study. This study is not blinded.

Subject type and number : The study population will be adults with unresectable locally advanced or metastatic solid tumors, whose disease has progressed despite standard therapy and for whom no further standard therapy exists; or for whom standard therapy has proven to be ineffective or intolerable.

This study is expected to enroll no more than 15 subjects, including malignant pleural mesothelioma and myxofibrosarcoma, 4-5, respectively, 2-3 malignant peripheral nerve sheath tumors, and other solid tumors.

Duration of treatment: Subjects will be treated with ES014 in 28-day cycles. ES014 will be administered at 1400 mg on days 1 and 15 of each cycle. Each subject will be treated with study drug for a maximum of 24 months. Subjects will be treated according to protocol until disease progression per RECIST v1.1, development of unacceptable toxicity, withdrawal of consent, completion of study treatment of 24 months, end of study, or early termination of study by sponsor, or other discontinuation and withdrawal reason, whichever occurs first.

DETAILED DESCRIPTION:
Subject type and number : The study population will be adults with unresectable locally advanced or metastatic solid tumors, whose disease has progressed despite standard therapy and for whom no further standard therapy exists; or for whom standard therapy has proven to be ineffective or intolerable.

* Cohort A: malignant pleural mesothelioma
* Cohort B: Mucinous fibrosarcoma
* Cohort C: Malignant peripheral nerve sheath tumour
* Cohort D: Other solid tumours

This study is expected to enroll no more than 15 subjects, including malignant pleural mesothelioma and myxofibrosarcoma, 4-5, respectively, 2-3 malignant peripheral nerve sheath tumors, and other solid tumors.

Duration of treatment: Subjects will be treated with ES014 in 28-day cycles. ES014 will be administered at 1400 mg on days 1 and 15 of each cycle. Each subject will be treated with study drug for a maximum of 24 months. Subjects will be treated according to protocol until disease progression per RECIST v1.1, development of unacceptable toxicity, withdrawal of consent, completion of study treatment of 24 months, end of study, or early termination of study by sponsor, or other discontinuation and withdrawal reason, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of unresectable locally advanced or metastatic solid tumours.
* Presence of at least one measurable lesion (according to RECIST v1.1).
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Life expectancy of at least 12 weeks.
* Adequate hematologic, hepatic, renal and coagulation functions per protocol.

Exclusion Criteria:

* Any prior therapy targeting CD39, CD73, adenosine A2A receptor, or TGF-β.
* Receipt of any investigational agents or devices within 4 weeks prior to the first dose of study drug.
* Prior treatment with the following therapies:

Anticancer therapy within 28 days or 5 half-lives of the drug prior to the first dose of study drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered with certain exceptions. A wash out of at least 2 weeks before the start of study drug for radiation to the extremities and 4 weeks for radiation to the chest, brain, or visceral organs is required.

* Prior allogeneic or autologous bone marrow transplant or solid organ transplant.
* Subject has received an infusion of blood products (including platelets or red blood cells), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), recombinant erythropoietin, or recombinant thrombopoietin within 14 days prior to the first administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the Efficacy of ES014 in Adult Subjects with Advanced Solid Tumours | 1-2 years
  ORR assessed by the investigators according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shuhang Wang, Ph.D, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China